CLINICAL TRIAL: NCT02202057
Title: Magnitude Estimation of Respiratory Resistive Load in Parkinson's Disease
Brief Title: Respiratory Load Magnitude Estimation in PD
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400183
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson's Disease; Aging
Keywords: respiratory sensation; somatosensation; resistive load; magnitude estimation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease: Men and women with Parkinson's disease, between 45 and 85 years of age. The following will be done: Respiratory resistive load on inhalation and Fluoroscopic swallowing evaluation.
  Interventions: Other: Respiratory resistive load on inhalation; Other: Fluoroscopic swallowing evaluation
- Healthy adults: Men and women without Parkinson's disease, between 45 and 85 years of age. The following will be done: Respiratory resistive load on inhalation.
  Interventions: Other: Respiratory resistive load on inhalation

INTERVENTIONS:
Other: Respiratory resistive load on inhalation — The participant will be seated in a chair, and will be instructed to "relax and breathe" through a facemask. Five respiratory resistive loads (5-40 cmH2O resistive pressure) will be applied between 3-5 times during inhalation. Following each loaded breath, participants will rate the perceived difficulty of breathing in.
Other: Fluoroscopic swallowing evaluation — Participants with PD only will receive a swallowing evaluation as part of their routine clinical care. Generally, the standard clinical evaluation protocol consists of multiple swallows of thin liquid barium, pudding-thick barium, and a cracker or cookie coated with barium. Results are reviewed by the treatment speech-language pathologist, and for the purposes of this study, the researchers will review the most recently recorded swallow study and identify the worst observed penetration-aspiration (PA) score.
  Groups: Parkinson's disease

SUMMARY:
The purpose of this study is to determine whether people with Parkinson's disease (PD) experience reduced perception of respiratory resistive loads versus healthy adults in the same age group. Further, the study will determine whether people with PD and trouble swallowing experience even more reduction of their perception of a respiratory resistive load.

DETAILED DESCRIPTION:
Experimental design and procedures: This prospective experimental study will be completed in one study visit taking between 1 and 3 hours. Verbal and written informed consent will be obtained by qualified members of the investigative team. Following informed consent, all participants will complete a health history questionnaire to assess inclusion/exclusion criteria. For patients with PD the consenting investigator will review the electronic medical record to ensure inclusion/exclusion criteria are met.

The experimental protocol will consist of 1.) Baseline pulmonary function measures, 2.) Baseline measures of depression and apathy, 3.) Presentation of resistive inspiratory loads via respiratory equipment, and 4.) Rating the perceived magnitude of respiratory sensations as measured on a modified Borg scale (ranging from 6 - no breathing difficulty - to 20 - maximal difficulty). For patients with PD only, the investigators will also review results of the rehabilitation barium swallow study performed as part of their standard clinical care.

Baseline Pulmonary function measures: The forced expired volume in the first second (FEV1) of a forced vital capacity (FVC) exhalation will be measured for each participant. Maximum inspiratory pressure (PiMax) will be measured with a manometer. The PiMax test will be repeated until 3 measurements within 10% variation are obtained, with at least 1 minute rest between trials.

Baseline depression and apathy: There is a significant impact for emotion on respiratory perceptual ratings. As such, we will measure baseline depression and apathy scores using 2 validated scales, the Beck Depression Index (BDI) and Marin Apathy Index (MAI). These are not outcome measures, but will be used to determine exclusion criteria.

Should depression (17 or greater on BDI) be detected in a participant, that participant will be provided with contact information for the University of Florida (UF) psychiatry and psychology clinic and encouraged to seek further evaluation. In the case severe depression is detected (31 or greater on BDI) the participant will not continue with the study, and will be provided with contact information for the UF psychiatry and psychology clinic and encouraged to seek further evaluation.

Inspiratory resistive load presentation:

The participant will be seated in a chair, separated from the investigator and experimental apparatus. The participant will be instructed to "relax and breathe" through a facemask connected to a non-rebreathing valve in line with a differential pressure transducer. The inspiratory port of the valve will be connected to the resistive loading manifold. The manifold consists of 5 differential resistors ranging from 5 - 40 centimeters/water (cmH2O) of resistive pressure, separated by stoppered ports, as well as a no load condition. The load is applied by removing the stop for an entire inspiratory breath, and then replacing the port to continue resting tidal breathing. The pressure transducer will provide measures of mouth pressure and airflow, which will be digitized and recorded to a desk top computer using LabChart software. Following each loaded breath, the participant will provide an estimate of the perceived difficulty of breathing using a modified Borg scale.

Participants will be familiarized with the loads in a practice session prior to initiating the experimental protocol. During the experimental session, participants will listen to music of their choice in order to mask experimental sounds. The resistive loads will be applied in a randomized block design, with each loaded breath separated by at least three unloaded breaths. Two blocks will be completed with each load presented between 3 and 5 times within each block. Therefore, there will be a total of between 15 and 25 loaded breaths (3-5 loads x 5 presentations) per block. Participants will be instructed that when they see a small light flash briefly on the table in front of them (which they will be familiarized with prior to beginning the experiment) a resistive load will be applied to the next breath. Following the loaded breath, the participant will be asked to estimate the perceived difficulty of breathing on the Borg scale.

Rehabilitation barium swallow study: Participants with PD who are referred for a rehabilitation barium swallowing evaluation will be recruited for this study. Therefore, the swallowing evaluation is part of the normal clinical care of the patients and may vary based on the clinical necessity as judged by the treating speech-language pathologist. Generally, the standard clinical evaluation protocol consists of multiple swallows of thin liquid barium, pudding-thick barium, and a cracker or cookie coated with barium. For the purposes of this study, the researchers will review the most recently recorded swallow study and identify the worst observed penetration-aspiration (PA) score (ranging from 1-8, where 1 is no penetration or aspiration, and 8 is silent aspiration). The PA score will be recorded in order to determine whether the participant has trouble swallowing (scores of 3-8) or not (scores of 1 and 2).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 45 and 85
* Ability to provide informed consent
* Patient group: Diagnosis of PD, Hoehn and Yahr stages II - IV, by a UF Movement Disorders fellowship trained neurologist having completed a clinical assessment of each participant's PD severity and arriving at the diagnosis of PD by applying strict UF brain bank criteria.
* Healthy older adults: History of PD, or any other neurologic or neurodegenerative disease including stroke.

Exclusion Criteria:

* History of head and neck cancer, and radiation treatment to the head or neck
* History of breathing disorders or diseases (e.g. chronic obstructive pulmonary disease (COPD), asthma, lung cancer)
* History of smoking in the past 5 years, or for more than 5 years at any one time
* Severe cognitive deficits including dementia.
* Difficulty complying with protocol due to severe neuropsychological disorder (i.e., severe depression: 31 or greater on the BDI)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 2 participant groups: those with Parkinson's disease, and healthy age- matched control participants. We will recruit 40 healthy older adults and 40 individuals with PD to participate. We will recruit all participants with PD from those referred for swallowing evaluation by the speech-language pathology service at the University of Florida (UF) Center for Movement Disorders and Neurorestoration (CMDNR). Healthy participants will be recruited via the UF Institutional Review Board's (IRBs) Healthstreet program, and local/campus advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Perceived difficulty inhaling against each respiratory resistive load. | Baseline
  Participants will rate the level of difficulty when inhaling against different levels of resistive load. The Borg scale ranges from 6-20, where 6 is 'no difficulty' and 20 is 'maximal difficulty.'

SECONDARY OUTCOMES:
The amount of pressure generated while inhaling against each resistive load | Baseline
  The mouth pressure will be measured while each participant is inhaling through the facemask, against each resistive load level. This will be measured in cmH2O

OTHER OUTCOMES:
Total amount of air that can be expired from the lungs | Baseline
  Spirometry will be used to determine the forced vital capacity, and forced expiratory volume in 1 second.
The maximum amount of inspiratory pressure | Baseline
  A manometer will be used to measure the maximum inspiratory pressure each participant can generate.
Feelings of sadness or depression | Baseline
  The Beck Depression Index (BDI) is a 21-item questionnaire that will be completed by each participant. Scores range from 1-10 (normal ups and downs) to over 40 (extreme depression).
Feeling apathetic, or indifferent. | Baseline
  The Marin apathy index (MAI) is a 14-item questionnaire with scores ranging from 0 (not at all) to 3 (a lot) for each item.
Ability to swallow liquids and solids without material entering the airway | Baseline
  The penetration-aspiration scale will be used by the investigators to determine whether material enters the airway during swallowing. This ranges from 1 (no penetration/aspiration) to 8 (silent aspiration).

CONTACTS AND LOCATIONS:
Overall Officials: Karen W Hegland, PHD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States